CLINICAL TRIAL: NCT00144469
Title: A Phase III Study of Ro25-8310 (Peginterferon Alfa-2a) in Combination With Ro20-9963 (Ribavirin) in Patients With Chronic Hepatitis C
Brief Title: A Study of Peginterferon Alfa-2a in Combination With Ribavirin in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JV15725
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: peginterferon alfa-2a
Drug: rivavirin

SUMMARY:
This study evaluated the efficacy and safety of the combination of peginterferon alfa-2a plus ribavirin in treatment-naïve patients with HCV genotype 1b infection, compared with peginterferon alfa-2a monotherapy.

Additionally, the study evaluated the efficacy and safety of the combination of peginterferon alfa-2a plus ribavirin in patients with CHC who had failed to respond to previous conventional-interferon based therapy.

DETAILED DESCRIPTION:
Treatment-naïve patients were randomly assigned in a 1:1 ratio to 48 weeks of double-blind treatment with subcutaneous, once-weekly injections of 180 μg of peginterferon alfa-2a (40KD) plus either twice-daily oral ribavirin (600 to 1000mg/day) or placebo.

All patients who had received previous treatment with conventional interferon but had failed to respond (no suppression of HCV-RNA below detection limits of a sensitive assay) or had relapsed (reversion to HCV-RNA positive state after suppression) received the combination of peginterferon alfa-2a (40KD) plus ribavirin for 48 weeks at the dosages stated above.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with quantifiable serum HCV-RNA (≥500 IU/mL))
* elevated serum alanine aminotransferase activity (≥45 IU per liter)within six months of screening
* liver biopsy findings consistent with a diagnosis of chronic hepatitis C.

Exclusion Criteria:

* Patients with neutropenia (fewer than 1,500 neutrophils per cubic millimeter)
* leukopenia (fewer than 3,000 white blood cells per cubic millimeter)
* thrombocytopenia (fewer than 90,000 platelets per cubic millimeter)
* anemia (less than 12 g hemoglobin per deciliter )
* hepatitis B co-infection
* decompensated liver disease
* organ transplant
* creatinine clearance less than 50 milliliters per minute
* poorly controlled psychiatric disease
* poorly controlled diabetes
* malignant neoplastic disease
* severe cardiac or chronic pulmonary disease
* immunologically mediated disease
* retinopathy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2002-05; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Sustained virological response, defined as undetectable HCV-RNA (<50IU per milliliter) after 24 weeks of untreated follow-up (week 72).

SECONDARY OUTCOMES:
Biochemical response (normalization of serum alanine aminotransferase activity),
Virological response (HCV-RNA <50IU per milliliter) at the end of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hirokazu Furuta, Study Director — Chugai Pharmaceutical